CLINICAL TRIAL: NCT04767282
Title: Innovative Nutrition Practices in Pediatric Health Care: Assessment of a Fruit and Vegetable Prescription Program for Children in Need
Brief Title: Assessment of a Fruit and Vegetable Prescription Program for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Hurley Medical Center (Other); Akpinar Children's Clinic (Unknown); Mott Children's Health Center (Other); Hurley Children's Center (Unknown)
Responsible Party: Principal Investigator, Amy Saxe-Custack, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003370; R01HD102527 (NIH)
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Exposure to Fruit and Vegetable Prescription Program
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Intervention Model Description: A fruit and vegetable prescription is written by pediatricians to exchange for $15 of fresh produce. Prescriptions are redeemable at a local farmers' market and mobile market.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruit and Vegetable Prescription (Other): Each program participant will receive a fruit and vegetable prescription that is written by pediatricians to exchange for $15 of fresh produce. Prescriptions will be distributed during pediatric office visits and are redeemable at a local farmers' market and mobile market.
  Interventions: Other: Fruit and Vegetable Prescription

INTERVENTIONS:
Other: Fruit and Vegetable Prescription — $15 voucher for fruit and vegetables

SUMMARY:
The objective of this study is to address gaps in knowledge related to the influence of pediatric fruit and vegetable prescription programs on food security, child dietary patterns, and weight status. To do this, we will compare demographically similar pediatric patient groups from three large clinics in a low-income urban city based on their exposure to a fruit and vegetable prescription program (FVPP) that provides one $15 prescription for fresh fruits and vegetable to every child at every office visit. Three clusters will be identified based on child exposure to the pediatric FVPP at baseline: high exposure (>24 months), moderate exposure (12-24 months), and no previous exposure. We will then introduce the FVPP to never exposed patients and collect, record, and compare changes in dietary intake, food security, and weight status over time. We will test the hypothesis that exposure to the FVPP is associated with higher intake of fruits and vegetables, better food security, and lower rates of obesity among children. The first aim will compare baseline dietary intake, food security, and weight status between high exposure, moderate exposure, no exposure groups. The second aim will measure changes in diet, food security, and weight status at 6-, 12-, 18-, and 24-months among children newly exposed to the FVPP. The third aim will compare follow-up measures of dietary intake, food security, and weight status in the initial no exposure group to baseline measures in the high exposure group.

DETAILED DESCRIPTION:
This study will evaluate a Fruit and Vegetable Prescription Program (FVPP). The program provides one $15 prescription for fresh produce to every child at every office visit. Prescriptions are redeemable at a local farmers' market and mobile market. To determine whether exposure to the FVPP is associated with improvements in dietary intake, food security, and health status, we will compare demographically similar pediatric patient groups with varying levels of exposure to the FVPP at baseline: high exposure (>24 months), moderate exposure (12-24 months), and no previous exposure. We will then introduce the FVPP to never exposed patients and collect, record, and compare changes in dietary intake, food security, and weight status over time. The central hypothesis is that exposure to the FVPP is associated with higher intake of fruits and vegetables, better food security, and lower rates of childhood obesity over time.

We propose the following three specific aims to test our hypothesis:

Aim 1 - Compare baseline dietary intake, food security, and weight status between pediatric patients with varying levels of exposure to the FVPP.

Aim 2 - Measure changes in diet, food security, and weight status when never exposed children are introduced to the FVPP.

Aim 3 - Compare mean follow-up measures of dietary intake, food security, and weight status in the initial no exposure group to baseline measures in the high exposure group.

ELIGIBILITY:
Inclusion Criteria:

* Child between age 8 and 16 years and their caregiver;
* Child active patient at clinic;
* Child received at least one fruit and vegetable prescription;
* Child and caregiver English-speaking

Exclusion Criteria:

* Caregiver or child not English speaking;
* Legal guardian not present at enrollment;
* Child assent refused;
* Sibling previously enrolled (one caregiver and one child per household);
* Movement between participating clinics

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Saxe-Custack, PhD, MPH, RD, Principal Investigator — Michigan State University
Locations (3):
- United States (3):
  - Hurley Children's Clinic, Flint, Michigan
  - Mott Children's Health Center, Flint, Michigan
  - Akpinar Children's Clinic, Flint, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Although the final dataset will be removed of identifiers prior to release for sharing, there remains the possibility of deductive disclosure of participants. Therefore, we will make all individual participant data that underlie results in publications available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Time Frame: Beginning 6 months after publication of final study results for a period of one year.
Access Criteria: Although the final dataset will be removed of identifiers prior to release for sharing, there remains the possibility of deductive disclosure of participants. Therefore, we will make all individual participant data that underlie results in publications available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Saxe-Custack A, Lofton HC, Hanna-Attisha M, Victor C, Reyes G, Ceja T, LaChance J. Caregiver perceptions of a fruit and vegetable prescription programme for low-income paediatric patients. Public Health Nutr. 2018 Sep;21(13):2497-2506. doi: 10.1017/S1368980018000964. Epub 2018 Apr 18. PMID 29667562
- [Background] Saxe-Custack A, LaChance J, Hanna-Attisha M, Ceja T. Fruit and Vegetable Prescriptions for Pediatric Patients Living in Flint, Michigan: A Cross-Sectional Study of Food Security and Dietary Patterns at Baseline. Nutrients. 2019 Jun 25;11(6):1423. doi: 10.3390/nu11061423. PMID 31242555
- [Background] Saxe-Custack A, LaChance J, Hanna-Attisha M. Child Consumption of Whole Fruit and Fruit Juice Following Six Months of Exposure to a Pediatric Fruit and Vegetable Prescription Program. Nutrients. 2019 Dec 20;12(1):25. doi: 10.3390/nu12010025. PMID 31877635
- [Background] Saxe-Custack A, Sadler R, LaChance J, Hanna-Attisha M, Ceja T. Participation in a Fruit and Vegetable Prescription Program for Pediatric Patients is Positively Associated with Farmers' Market Shopping. Int J Environ Res Public Health. 2020 Jun 12;17(12):4202. doi: 10.3390/ijerph17124202. PMID 32545578
- [Background] Saxe-Custack A, Todem D, Anthony JC, Kerver JM, LaChance J, Hanna-Attisha M. Effect of a pediatric fruit and vegetable prescription program on child dietary patterns, food security, and weight status: a study protocol. BMC Public Health. 2022 Jan 21;22(1):150. doi: 10.1186/s12889-022-12544-y. PMID 35062926
- [Background] Saxe-Custack A, Egan S, Farmer B, Pulka K, Sampson A. Caregiver-reported barriers to engagement in a paediatric fresh fruit and vegetable prescription programme. J Nutr Sci. 2024 Sep 18;13:e33. doi: 10.1017/jns.2024.33. eCollection 2024. PMID 39314532
- [Result] Saxe-Custack A, Todem D, LaChance J, Kerver J, Anthony J. Association between youth blood pressure and exposure to pediatric fruit and vegetable prescriptions. Pediatr Res. 2025 Aug;98(2):654-662. doi: 10.1038/s41390-024-03671-w. Epub 2024 Dec 10. PMID 39653792
- [Result] Sadler RC, Saxe-Custack A. 'Nobody Shops at the Neighborhood Store': Leveraging a Community's Pediatric Fresh Produce Prescription Program to Inform Future Participating Store Redemption Locations. Cities Health. 2024;8(1):70-81. doi: 10.1080/23748834.2023.2281764. Epub 2023 Nov 23. PMID 38585045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregiver-child dyads were recruited from February 2021 through June 2022 at pediatric clinics in Flint, Michigan. The high exposure clinic is a large pediatric clinic that introduced Michigan's first pediatric fruit and vegetable prescription program in February 2016. The moderate exposure clinic is one of the largest private-practice pediatric clinics in Flint serving over 3,000 patients. The no/low exposure clinic is the largest pediatric clinic in Flint.
Pre-assignment Details: Exposure to the pediatric fruit and vegetable prescription program was based on length of time a child was a patient at one of three partnering clinics that offered the fruit and vegetable prescription program. Number of participants started represents the number of individual participants (caregivers and children).
Groups:
- Moderate Exposure to the FVPP: Patients with Moderate Exposure to the FVPP
- High Exposure to the FVPP: Patients with High Exposure to the FVPP
- No/Low Exposure to the FVPP: Patients with No/Low Exposure to the FVPP
Period: Overall Study
Arm/Group | Moderate Exposure to the FVPP | High Exposure to the FVPP | No/Low Exposure to the FVPP
Started | 362 | 406 | 632
Children | 181 | 203 | 316
Caregivers | 181 | 203 | 316
Completed | 350 | 402 | 608
Not Completed | 12 | 4 | 24
Not completed — Refused or did not begin surveys | 6 | 2 | 2
Not completed — Duplicate household previously enrolled | 2 | 0 | 8
Not completed — Unable to confirm legal guardian | 0 | 2 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 6
Not completed — Survey comprehension challenges | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate Exposure to the FVPP: Participants with Moderate Exposure to the FVPP
- High Exposure to the FVPP: Participants with High Exposure to the FVPP
- No/Low Expsoure to the FVPP: Participants with No/Low Exposure to the FVPP
- Total: Total of all reporting groups
Arm/Group | Moderate Exposure to the FVPP | High Exposure to the FVPP | No/Low Expsoure to the FVPP | Total
Number analyzed (Participants) | 350 | 402 | 608 | 1360
Age, Categorical [Count of Participants; unit: Participants] — Population: For the age distribution, 11 participants did not provide their age. So, 1349 participants did provide data to generate the age at enrollment.
  Participants
    number analyzed (Participants) | 348 | 402 | 599 | 1349
    <=18 years | 175 | 201 | 300 | 676
    Between 18 and 65 years | 167 | 198 | 291 | 656
    >=65 years | 6 | 3 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: For the age distribution, 11 participants did not provide their age. So, 1349 participants did provide data to generate the age at enrollment.
  years
    Age: number analyzed (Participants) | 348 | 402 | 599 | 1349
    Age | 26.99 (15.61) | 25.92 (14.87) | 25.72 (15.54) | 26.11 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For the sex distribution, 4 participants did not provide their sex. So, 1356 participants did provide data on their sex modality. Additionally, the number analyzed in row differs from overall because the first row (titled Total) represents the overall study sample (children and caregivers).
  Participants
    Total: number analyzed (Participants) | 350 | 402 | 604 | 1356
    Total: Female | 250 | 282 | 428 | 960
    Total: Male | 100 | 120 | 176 | 396
    Children: number analyzed (Participants) | 175 | 201 | 304 | 680
    Children: Female | 91 | 103 | 159 | 353
    Children: Male | 84 | 98 | 145 | 327
    Caregivers: number analyzed (Participants) | 175 | 201 | 300 | 676
    Caregivers: Female | 159 | 179 | 269 | 607
    Caregivers: Male | 16 | 22 | 31 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number analyzed in row differs from overall because the first row (titled Total) represents the overall study sample (children and caregivers).
  Participants
    Total: Hispanic or Latino | 5 | 1 | 12 | 18
    Total: Not Hispanic or Latino | 341 | 401 | 579 | 1321
    Total: Unknown or Not Reported | 4 | 0 | 17 | 21
    Children: number analyzed (Participants) | 175 | 201 | 304 | 680
    Children: Hispanic or Latino | 2 | 0 | 5 | 7
    Children: Not Hispanic or Latino | 172 | 201 | 289 | 662
    Children: Unknown or Not Reported | 1 | 0 | 10 | 11
    Caregivers: number analyzed (Participants) | 175 | 201 | 304 | 680
    Caregivers: Hispanic or Latino | 3 | 1 | 7 | 11
    Caregivers: Not Hispanic or Latino | 169 | 200 | 290 | 659
    Caregivers: Unknown or Not Reported | 3 | 0 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total in subgroups does not include Hispanics. There are 5, 1 and 12 Hispanics in high, moderate and no/low exposure group respectively. Additionally, the number analyzed in row differs from overall because the first row (titled Total) represents the overall study sample (children and caregivers).
  Participants
    Total: number analyzed (Participants) | 345 | 401 | 596 | 1342
    Total: American Indian or Alaska Native | 3 | 5 | 3 | 11
    Total: Asian | 1 | 2 | 4 | 7
    Total: Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
    Total: Black or African American | 253 | 330 | 414 | 997
    Total: White | 68 | 47 | 129 | 244
    Total: More than one race | 15 | 17 | 27 | 59
    Total: Unknown or Not Reported | 4 | 0 | 17 | 21
    Children: number analyzed (Participants) | 173 | 201 | 299 | 673
    Children: American Indian or Alaska Native | 1 | 3 | 2 | 6
    Children: Asian | 1 | 1 | 1 | 3
    Children: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
    Children: Black or African American | 128 | 165 | 212 | 505
    Children: White | 30 | 19 | 57 | 106
    Children: More than one race | 11 | 13 | 16 | 40
    Children: Unknown or Not Reported | 1 | 0 | 10 | 11
    Caregivers: number analyzed (Participants) | 172 | 200 | 297 | 669
    Caregivers: American Indian or Alaska Native | 2 | 2 | 1 | 5
    Caregivers: Asian | 0 | 1 | 3 | 4
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    Caregivers: Black or African American | 125 | 165 | 202 | 492
    Caregivers: White | 38 | 28 | 72 | 138
    Caregivers: More than one race | 4 | 4 | 11 | 19
    Caregivers: Unknown or Not Reported | 3 | 0 | 7 | 10
Region of Enrollment [Number; unit: participants]
  United States | 350 | 402 | 608 | 1360
Age of Study Participants [Mean (Standard Deviation); unit: Years] — Population: There were missing data either with the youth or adult data.
  Years
    Age of youth participants: number analyzed (Participants) | 175 | 201 | 300 | 676
    Age of youth participants | 12.93 (2.34) | 12.47 (2.63) | 11.98 (2.39) | 12.37 (2.48)
    Age of adult participants: number analyzed (Participants) | 173 | 201 | 299 | 673
    Age of adult participants | 41.22 (9.02) | 39.74 (8.53) | 39.51 (9.89) | 39.91 (9.30)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Child-reported Mean Daily Intake of Fruits and Vegetables at 6 and 12 Months Among Youth Participants Newly Introduced to the FVPP
Description: Eating behaviors reported here were assessed via child-report using the 41-item Block Kids Food Screener (BKFS), chosen for low respondent burden and acceptable psychometric values. Dietary analysis, using Block Online Analysis System, provided nutrient estimates and number of servings by food groups. This data was used to determine mean daily intake (in cup equivalents) of total vegetables, total fruits, and whole fruits.
Time Frame: Baseline, 6 months,12 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" group. Analysis includes data from youth participants with no/low exposure to the FVPP at baseline who completed the Block Kids Food Screener.
Measure: Mean (95% Confidence Interval); unit: cup equivalents per day
Groups:
- No/Low Exposure: Patients with the lowest exposure to the pediatric fruit and vegetable prescription program at baseline who were followed for 24 months to assess changes in outcome measures.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 300
cup equivalents per day
  Change in mean daily intake of total fruits (6 months versus baseline) | 0.21 [0.00 to 0.41]
  Change in mean daily intake of total fruits (12 months versus baseline) | 0.17 [-0.01 to 0.34]
  Change in mean daily intake of whole fruits (6 months versus baseline) | 0.14 [0.01 to 0.26]
  Change in mean daily intake of whole fruits (12 months versus baseline) | 0.05 [-0.06 to 0.16]
  Change in mean daily intake of total vegetables (6 months versus baseline) | 0.11 [-0.06 to 0.28]
  Change in mean daily intake of total vegetables (12 months versus baseline) | -0.01 [-0.14 to 0.12]

2. Primary Outcome: Odds Ratio Evaluating the Longitudinal Trend of High Food Security for the Household at 6 and 12 Months Relative to Baseline Among Caregivers Newly Introduced to the FVPP
Description: Household food security was assessed using the US Household Food Security Module: Six Item Short Form (National Center for Health Statistics) via caregiver report. The sum of affirmative responses to six questions served as the household's raw score. Food security status was assigned based on a calculated raw score (0-1=high/marginal food security; 2-4=low food security; 5-6 very low food security). High food security (outcome analyzed) was assigned to those with raw scores less than or equal to 1.
Time Frame: Baseline, 6 months,12 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" group. Analysis includes data from caregivers with no/low exposure to th FVPP at baseline who completed the entire US Household Food Security Module.
Measure: Number (95% Confidence Interval); unit: High Food Security Odds Ratio
Groups:
- No/Low Exposure: Patients with the lowest exposure to the pediatric fruit and vegetable prescription program at baseline.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 300
High Food Security Odds Ratio
  Odds ratios for higher food security (6 months versus baseline) | 0.87 [0.59 to 1.29]
  Odds ratios for higher food security (12 months versus baseline) | 0.92 [0.61 to 1.37]

3. Primary Outcome: Odds Ratio Evaluating the Longitudinal Trend of High Food Security at 6 and 12 Months Relative to Baseline Among Youth 12 Years of Age and Older Who Were Newly Introduced to the FVPP.
Description: Child food security status was assessed via the Self-Administered Food Security Survey Module for Youth only with children aged 12 years and older based on prior research recommendations. The sum of affirmative responses ("a lot" or "sometimes") to nine questions represented the respondent's raw score on the scale. Food security status was assigned by raw score (0-1=high/marginal food security; 2-5=low food security; 6-9=very low food security). High food security (outcome analyzed) was assigned to those with raw scores less than or equal to 1.
Time Frame: Baseline, 6 months,12 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" group. Analysis includes data from youth 12 years of age and older who were newly introduced to the FVPP and completed the Self-Administered Food Security Survey Module for Youth.
Measure: Number (95% Confidence Interval); unit: High Food Security Odds Ratio
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 142
High Food Security Odds Ratio
  Odds ratios for higher food security (6 months versus baseline) | 0.86 [0.39 to 1.90]
  Odds ratios for higher food security (12 months versus baseline) | 0.64 [0.32 to 1.28]

4. Primary Outcome: Odds Ratio Evaluating the Longitudinal Trend of High Food Security at 6, 12, 18 and 24 Months Relative to Baseline Among Youth 12 Years of Age and Older at Newly Introduced to the FVPP
Description: as for outcome 3
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: High Food Security Odds Ratio
Groups:
- No/Low Exposure: Patients with the lowest exposure to the pediatric fruit and vegetable prescription program at baseline and were followed for 24 months to assess changes in outcome measures.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 142
High Food Security Odds Ratio
  Odds ratios for higher food security (6 months versus baseline) | 0.86 [0.39 to 1.90]
  Odds ratios for higher food security (12 months versus baseline) | 0.64 [0.32 to 1.28]
  Odds ratios for higher food security (18 months versus baseline) | 0.48 [0.25 to 0.95]
  Odds ratios for higher food security (24 months versus baseline) | 0.39 [0.19 to 0.78]

5. Primary Outcome: Change From Baseline Child-reported Mean Daily Intake of Fruits and Vegetables at 6, 12, 18 and 24 Months Among Youth Participants Newly Introduced to the FVPP
Description: as for outcome 1
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" groups. Analysis includes data from youth participants who were newly introduced to the FVPP and completed the Block Kids Food Screener.
Measure: Mean (95% Confidence Interval); unit: cup equivalents per day
Groups:
- No/Low Exposure: Patients with the lowest baseline exposure to the pediatric fruit and vegetable prescription program who were followed for 24 months to assess changes in outcome measures.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 300
cup equivalents per day
  Change in mean daily intake of total fruits (6 months versus baseline) | 0.21 [0.00 to 0.41]
  Change in mean daily intake of total fruits (12 months versus baseline) | 0.17 [-0.01 to 0.34]
  Change in mean daily intake of total fruits (18 months versus baseline) | 0.37 [0.19 to 0.55]
  Change in mean daily intake of total fruits (24 months versus baseline) | 0.09 [-0.10 to 0.29]
  Change in mean daily intake of whole fruits (6 months versus baseline) | 0.14 [0.01 to 0.26]
  Change in mean daily intake of whole fruits (12 months versus baseline) | 0.05 [-0.06 to 0.16]
  Change in mean daily intake of whole fruits (18 months versus baseline) | 0.20 [0.09 to 0.32]
  Change in mean daily intake of whole fruits (24 months versus baseline) | 0.12 [-0.00 to 0.25]
  Change in mean daily intake of total vegetables (6 months versus baseline) | 0.11 [-0.06 to 0.28]
  Change in mean daily intake of total vegetables (12 months versus baseline) | -0.01 [-0.14 to 0.12]
  Change in mean daily intake of total vegetables (18 months versus baseline) | 0.19 [0.03 to 0.35]
  Change in mean daily intake of total vegetables (24 months versus baseline) | -0.02 [-0.16 to 0.12]

6. Primary Outcome: Odds Ratio Evaluating the Longitudinal Trend of High Food Security for the Household at 6, 12, 18 and 24 Months Relative to Baseline Among Caregivers Newly Introduced to the FVPP
Description: as for outcome 2
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" group. Analysis includes data from caregivers newly introduced to the FVPP who completed the US Household Food Security Module.
Measure: Number (95% Confidence Interval); unit: High Food Security Odds Ratio
Groups:
- No/Low Exposure: Patients with the lowest exposure to the pediatric fruit and vegetable prescription program who were followed for 24 months to assess changes in outcome measures.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 300
High Food Security Odds Ratio
  Odds ratios for higher food security (6 months versus baseline) | 0.87 [0.59 to 1.29]
  Odds ratios for higher food security (12 months versus baseline) | 0.92 [0.61 to 1.37]
  Odds ratios for higher food security (18 months versus baseline) | 0.71 [0.47 to 1.07]
  Odds ratios for higher food security (24 months versus baseline) | 0.92 [0.59 to 1.46]

7. Secondary Outcome: Change From Baseline Child BMI at 6 and 12 Months Among Youth Participants Newly Introduced to the FVPP
Description: Body mass index (BMI) was calculated from child weight and height (weight (kg)/[height (m)]2). BMI was then categorized into percentiles by sex and age to serve as an indicator of overweight and obesity. Child overweight and obesity status were categorized as follows: overweight (95th percentile for age and sex > BMI ≥ 85th percentile for age and sex), obese (BMI ≥ 95th percentile for age and sex). Because achievement of healthy weight in youth (85th percentile for age and sex ≥ BMI > 5th percentile for age and sex) was a secondary objective, a negative change in BMI percentile represents a desirable outcome.
Time Frame: Baseline, 6 months,12 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" group. Pediatric patients with recorded height and weight measurements.
Measure: Mean (95% Confidence Interval); unit: BMI percentile
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 296
BMI percentile
  Change in BMI percentiles (6 months versus baseline) | -0.48 [-2.46 to 1.50]
  Change in BMI percentile (12 months versus baseline) | -1.93 [-3.36 to -0.50]

8. Secondary Outcome: Change From Baseline BMI at 6, 12, 18 and 24 Months Among Youth Participants Newly Introduced to the FVPP
Description: as for outcome 7
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: BMI percentile
Groups:
- No/Low Exposure: Patients had the lowest exposure to the pediatric fruit and vegetable prescription program at baseline and were followed for 24 months to assess changes in outcome measures.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 296
BMI percentile
  Change in BMI percentile (6 months versus baseline) | -0.48 [-2.46 to 1.50]
  Change in BMI percentile (12 months versus baseline) | -1.93 [-3.36 to -0.50]
  Change in BMI percentile (18 months versus baseline) | -1.98 [-3.88 to -0.08]
  Change in BMI percentile (24 months versus baseline) | -3.43 [-5.30 to -1.57]

9. Secondary Outcome: Change From Caregiver-reported Baseline Mean Daily Intake of Fruits and Vegetables at 6 and 12 Months Among Caregivers Newly Introduced to the FVPP
Description: To investigate whether exposure to the pediatric fruit and vegetable prescription program is associated with increased fruit and vegetable consumption among caregivers, dietary data from caregivers was collected using the National Cancer Institute Fruit & Vegetable Intake "All Day" Screener which asks frequency and portion size questions about nine food items. This will be used to calculate mean daily intake of vegetables and total fruits.
Time Frame: Baseline, 6 months, 12 months
Population: This outcome measure was pre-specified to only assess participants in the "low/no exposure to FVPP" group. Analysis includes data from caregivers newly introduced to the FVPP who completed the NCI All Day Screener.
Measure: Mean (95% Confidence Interval); unit: cup equivalents per day
Groups:
- No/Low Exposure: Patients had the lowest exposure to the pediatric fruit and vegetable prescription program at baseline.
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 299
cup equivalents per day
  Change in mean daily intake of fruits and vegetables (6 months versus baseline) | -0.21 [-1.00 to 0.58]
  Change in mean daily intake of fruits and vegetables (12 months versus baseline) | -0.56 [-1.14 to 0.01]

10. Secondary Outcome: Change From Caregiver-reported Baseline Mean Daily Intake of Fruits and Vegetables at 6, 12, 18 and 24 Months Among Caregivers Newly Introduced to the FVPP
Description: as for outcome 9
Time Frame: Baseline, 6 months, 12 months, 18 months, 24 months
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: cup equivalents per day
Arm/Group | No/Low Exposure
Number analyzed (Participants) | 299
cup equivalents per day
  Change in mean daily intake of fruits and vegetables (6 months versus baseline) | -0.21 [-1.00 to 0.58]
  Change in mean daily intake of fruits and vegetables (12 months versus baseline) | -0.56 [-1.14 to 0.01]
  Change in mean daily intake of fruits and vegetables (18 months versus baseline) | -0.90 [-1.73 to -0.07]
  Change in mean daily intake of fruits and vegetables (24 months versus baseline) | -0.50 [-1.08 to 0.09]

ADVERSE EVENTS:
Time Frame: 3 Years
Groups:
- All Participants: All study participants
- Children With High Exposure to the FVPP: Pediatric Patients with High Exposure to the FVPP
- Caregivers With High Expsoure to the FVPP: Caregivers of Pediatric Patients with High Exposure to the FVPP
- Children With Moderate Exposure to the FVPP: Pediatric Patients with Moderate Exposure to the FVPP
- Caregivers With Moderate Exposure to the FVPP: Caregivers of Pediatric Patients with Moderate Exposure to the FVPP
- Children With No/Low Exposure to the FVPP: Pediatric Patients with No/Low Exposure to the FVPP
- Caregivers With No/Low Exposure to the FVPP: Caregivers of Pediatric Patients with No/Low Exposure to the FVPP
Arm/Group | All Participants | Children With High Exposure to the FVPP | Caregivers With High Expsoure to the FVPP | Children With Moderate Exposure to the FVPP | Caregivers With Moderate Exposure to the FVPP | Children With No/Low Exposure to the FVPP | Caregivers With No/Low Exposure to the FVPP
All-Cause Mortality (participants affected / at risk) | 0/1360 | 0/201 | 0/201 | 0/175 | 0/175 | 0/304 | 0/304
Serious Adverse Events (participants affected / at risk) | 0/1360 | 0/201 | 0/201 | 0/175 | 0/175 | 0/304 | 0/304
Other Adverse Events (participants affected / at risk) | 0/1360 | 0/201 | 0/201 | 0/175 | 0/175 | 0/304 | 0/304

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT04767282/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT04767282/ICF_000.pdf